CLINICAL TRIAL: NCT02367313
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Dose-ranging Study of Vapendavir in Moderate to Severe Asthmatic Adults With Symptomatic Human Rhinovirus Infection
Brief Title: A Phase 2 Study of Vapendavir in Asthmatic Adults With Symptomatic Human Rhinovirus Infection
Acronym: SPIRITUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biota Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA798-203; 2014-001785-95 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Symptomatic Human Rhinovirus Infection; Moderate to Severe Asthma; Antiviral; Cold; Aviragen Therapeutics, Inc.; Aviragen Therapeutics; Aviragen
MeSH Terms: conditions — Asthma; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Vapendavir 264 mg (Active Comparator): Vapendavir 264 mg and matching placebo
  Interventions: Drug: Vapendavir
- Vapendavir 528 mg (Active Comparator): Vapendavir 528 mg and matching placebo
  Interventions: Drug: Vapendavir

INTERVENTIONS:
Drug: Vapendavir — Vapendavir 264 mg twice daily
  Other Names: BTA798
  Arms: Vapendavir 264 mg
Drug: Vapendavir — Vapendavir 528 mg twice daily
  Other Names: BTA798
  Arms: Vapendavir 528 mg
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
This Phase 2 protocol is designed to compare two dose levels of Vapendavir versus placebo. The objectives are to obtain safety and efficacy data in moderate to severe asthmatic patients, aged 18 to 75 years at risk of loss of asthma control due to presumptive Human Rhinovirus infection.

DETAILED DESCRIPTION:
This is a multicenter trial to be conducted at approximately 60 sites among 6-8 northern hemisphere countries in North America and Central Europe. Sufficient patients will be randomized in order to recruit 150 subjects who are laboratory confirmed for human rhinovirus (HRV) infection. Depending on HRV PCR positivity rates, it is expected that randomization of 250-480 subjects will be required to achieve this number of subjects with HRV infection.

Appropriate asthma subjects will be screened up to 180 days prior to presentation at the study site with symptoms of presumed HRV infection for potential study inclusion on Study Day 1. The study drug treatment period has a duration of 7 days, beginning on Study Day 1. Follow-up study visits to the clinic occur on Study Days 3, 5, 7, 14, 21, and 28 with a telephonic final safety follow-up visit conducted on Study Day 35. Thus, depending on the duration of the screening period, a subject's duration of participation can be estimated to last from approximately 37 days up to 215 days.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate and severe male and female asthma subjects aged 18 to 75 years, (inclusive)
2. Established clinical history of Asthma for at least 1 year, and a history within the last 14 months (prior to screening) of asthma exacerbation due to presumed viral respiratory infections, which required asthma rescue medication treatment.
3. The asthma subjects will be currently taking at least medium-dose or high-dose ICS defined as fluticasone at a dosage of at least >264 µg daily and may be taking other asthma medication preparations. The asthma subjects' medication regimen must be stable for at least 4 weeks before screening.
4. Subjects will have at screening or within the last year, documented variable airway obstruction as indicated by an increase in FEV1 (>12%) to short acting bronchodilator, or positive methacholine challenge, or positive histamine challenge (PC20 <8 mg/mL).
5. Upon presentation to the clinic with cold symptoms, subjects will be required to be randomized and treated within 48 hours of symptom onset and will be qualified for presumptive rhinovirus infection by:

   1. clinical exam and the presence of each of the following Day 1 WURSS-21 symptoms at a severity of 2 or greater: runny nose, sore throat, scratchy throat.
   2. subjects must also have a minimum total symptom score on the Day 1 WURSS-21 of 20 points.
   3. subjects will be further qualified as presumptively infected with HRV via exclusion of subjects having significant fever and exclusion of subjects testing positive for influenza via Rapid Antigen Test.

Exclusion Criteria:

1. Subjects presenting to the clinic with a current severe asthma exacerbation will be excluded from randomization, as well as any subject with an additional underlying respiratory medical condition other than asthma such as COPD, cystic fibrosis, or chronic sinusitis, or any other uncontrolled clinically significant disease which would interfere with the assessment outcomes or subject safety.
2. Female subjects must not be pregnant or breastfeeding. Females of childbearing potential must be willing to utilize a double barrier method of contraception, as defined in this protocol, regardless of any hormonal contraception they may be concomitantly receiving.
3. Male subjects must agree to use a method of birth control defined in this protocol.
4. The use of medications known to moderately or severely inhibit or induce cytochrome (CYP) 3A4 and 2C19 enzymes, or those known to be sensitive substrates (with a narrow therapeutic range) of these CYPs are restricted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire-6 (ACQ-6) | Baseline (Day 1) to Study Day 14
  Least Square (LS) mean change from baseline (Day 1) to Study Day 14 in ACQ-6 total score

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Biota Pharmaceuticals, Inc.
Locations (56):
- United States (33):
  - Biota Investigational site, Birmingham, Alabama
  - Biota Investigational site, Flagstaff, Arizona
  - Biota Investigational site, Bakersfield, California
  - Biota Investigational site, Los Angeles, California
  - Biota Investigational site, Orange, California
  - Biota Investigational Site, San Jose, California
  - Biota Investigational site, Stockton, California
  - Biota Investigational site, Centennial, Colorado
  - Biota Investigational site, Denver, Colorado
  - Biota Investigational site, Hialeah, Florida
  - Biota Investigational site, New Port Richey, Florida
  - Biota Investigational site, Oviedo, Florida
  - Biota Investigation site, Palmetto Bay, Florida
  - Biota Investigational site, Tallahassee, Florida
  - Biota Investigational site, Twin Falls, Idaho
  - Biota Investigational site, Baltimore, Maryland
  - Biota Investigational site, St Louis, Missouri
  - Biota Investigational site, Bellevue, Nebraska
  - Biota investigational site, Las Vegas, Nevada
  - Biota Investigational site, Ocean City, New Jersey
  - Biota Investigational site, Albuquerque, New Mexico
  - Biota Investigational site, Rockville Centre, New York
  - Biota Investigational site, Raleigh, North Carolina
  - Biota Investigational site, Fargo, North Dakota
  - Biota Investigational site, Middleburg, Ohio
  - Biota Investigational site, Toledo, Ohio
  - Biota Investigation site, Oklahoma City, Oklahoma
  - Biota Investigational site, Medford, Oregon
  - Biota Investigational site, Portland, Oregon
  - Biota Investigational site, Warwick, Rhode Island
  - Biota Investigational site, Houston, Texas
  - Biota Investigational site, Seattle, Washington
  - Biota Investigational site, Greenfield, Wisconsin
- Bulgaria (3):
  - Biota Investigational site, Rousse
  - Biota Investigational site, Sofia
  - Biota Investigational site, Stara Zagora
- Czechia (6):
  - Biota Investigational site, Jindřichův Hradec
  - Biota Investigational site, Kyjov
  - Biota Investigational site, Lovosice
  - Biota Investigational site, Mělník
  - Biota Investigational site, Prague
  - Biota Investigational site, Rokycany
- Biota Investigational site, Tbilisi, Georgia
- Poland (8):
  - Biota Investigational site, Bialystok
  - Biota Investigational site, Kielce
  - Biota Investigational site, Krakow
  - Biota Investigational site, Lodz
  - Biota Investigational site, Lublin
  - Biota Investigational site, Skierniewice
  - Biota Investigational site, Warsaw
  - Biota Investigational site, Wroclaw
- Romania (5):
  - Biota Investigational site, Brasov
  - Biota Investigational site, Bucharest
  - Biota Investigational site, Craiova
  - Biota Investigational site, Mures
  - Biota Investigational site, Sibiu